CLINICAL TRIAL: NCT00774969
Title: Phase 1 Study to Evaluate the Pharmacokinetics of Metronidazole 10% Ointment Applied Peri-Anally in Healthy Volunteers and Patients With Perianal Crohn's Disease
Brief Title: Evaluation of the Pharmacokinetics of Metronidazole 10% Ointment Applied Peri Anally in Healthy Volunteers and Patients With Perianal Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: MET/PK/01; EudraCT/IND 2007003173-68
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Perianal Crohns'
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All (Experimental): 6 patients with Perianal Crohn's Disease and 10 healthy Volunteers
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Metronidazole 10% ointment three times a day 7 days

SUMMARY:
The purpose of this study is to evaluate the blood levels of Metronidazole after application to the peri anal area after a single dose and 6 or 7 days application.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Male and female patients with Crohn's disease (diagnosed by radiology, endoscopy and pathology), with anorectal involvement.
* Aged 18-65 years.
* Have had perianal symptoms for longer than 2 months
* Have a score of 5 or above in the Perianal Crohn's Disease Activity Index (PCDAI)
* Have a score of 1 or above on the 'Type of perianal disease' assessment of the PCDAI
* Subjects can be on concomitant medication. Acceptable regimens are:

  * Aminosalicylates at a dosage that has been stable for more than 4 weeks before screening;Infliximab on a stable infusion regimen;
  * Oral corticosteroids <40mg per day; Methotrexate, provided that dosage has been stable for more than 4 weeks; azathioprine or mercaptopurine at a dosage that has been stable for more than 8 weeks;
  * Antibiotics at a dosage that has been stable for 4 weeks but excluding metronidazole.
  * Cyclosporin on a stable dose for more than 4 weeks.
* If patients have setons these must have been in place for at least 4 weeks prior to screening.
* If female, the subject must not be lactating and must be (a) post-menopausal, (b) surgically sterilised, or (c) have a negative pregnancy test result prior to entry into the study and will use double-barrier methods of contraception (two separate methods of birth control, one of which may include oral contraception) for the duration of the study.
* Must have provided written informed consent to participate.

Healthy volunteer group:

* They have had surgery to the anus or rectum in the past 4 weeks.
* Have a history of inflammatory bowel disease.
* Allergic to metronidazole.
* Are taking any prohibited medication.
* Not prepared to refrain from drinking alcohol during the course of the study.
* Deemed mentally incompetent.
* Considered by their physician unlikely to be able to comply with the protocol.
* Has donated blood within the past 3 months.
* Taken part in an experimental drug study in the preceding three months.

Exclusion Criteria:

Patient group:

* They have had surgery to the anus or rectum in the past 4 weeks.
* They have a perianal abscess requiring incision and drainage.
* They have a stoma of less than 6 months duration.
* Allergic to metronidazole.
* Are taking any prohibited medication.
* Not prepared to refrain from drinking alcohol during the course of the study.
* Deemed mentally incompetent.
* Considered by their physician unlikely to be able to comply with the protocol.
* Has donated blood within the past 3 months.
* Taken part in an experimental drug study in the preceding three months.
* Has donated blood within the past 3 months.
* Taken part in an experimental drug study in the preceding three months.

Healthy volunteer group:

* They have had surgery to the anus or rectum in the past 4 weeks.
* Have a history of inflammatory bowel disease.
* Allergic to metronidazole.
* Are taking any prohibited medication.
* Not prepared to refrain from drinking alcohol during the course of the study.
* Deemed mentally incompetent.
* Considered by their physician unlikely to be able to comply with the protocol.
* Has donated blood within the past 3 months.
* Taken part in an experimental drug study in the preceding three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Jordan, BSC, Study Director — SLA Pharma
Locations (1):
- Sainsbury Wing, St Marks & Northwick Park Hospitals, Watford Road, Harrow, United Kingdom